CLINICAL TRIAL: NCT02133001
Title: A Double-blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Subjects Who Are Assessed to be at Imminent Risk for Suicide
Brief Title: A Double-blind Study to Assess the Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Participants Who Are Assessed to be at Imminent Risk for Suicide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103162; ESKETINSUI2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Esketamine; Intranasal esketamine; Placebo
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Esketamine (Experimental): Esketamine hydrochloride solution (containing 14 milligram (mg) of esketamine base per 100 microliter [mcl] of intranasal spray) will be administered by intranasal route using nasal spray pump as two times a week, for 4 weeks. Dose may be reduced to 56 mg per day based on Investigator's discretion.
  Interventions: Drug: Esketamine
- Placebo (Placebo Comparator): Matching Placebo solution will be administered by intranasal route using nasal spray pump as two times a week, for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — Esketamine 84 mg will be self-administered by participants as intranasal spray as two times a week, for 4 weeks (that is, Day 1,4,8,11,15,18,22,25). Dose may be reduced to 56 mg per day based on Investigator's discretion.
  Other Names: Esketamine hydrochloride
  Arms: Esketamine
Drug: Placebo — Matching placebo will be self-administered by participants as intranasal spray as two times a week, for 4 weeks (that is, Day 1,4,8,11,15,18,22,25).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of intranasal esketamine 84 milligram (mg) compared with intranasal placebo along with standard care treatment, in reducing the symptoms of major depressive disorder (MDD) (an affective disorder manifested by either a dysphoric mood or loss of interest or pleasure in usual activities, the mood disturbance is prominent and relatively persistent), including the risk for suicide as assessed by the Investigator, in participants who will be assessed to be at imminent risk for suicide.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither physician nor participant knows assigned study treatment), placebo-controlled (participants are randomly assigned to a test treatment or to an identical-appearing treatment that does not contain the test drug), and multicenter (when more than one hospital or medical school team works on a medical research study), study of esketamine in participants with major depressive disorder (MDD) in participants who will be assessed to be at imminent risk for suicide, as measured by the change from Baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) total score at 4 hours postdose on Day 1. The duration of study will be approximately 81 days per participant. The study consists of 3 parts: Screening (that is, with in 1 day before study commences on Day 1) and double-blind Treatment (from Day 1-25) and Follow-up (from Day 26 up to Day 81). All the eligible participants will be provided standard care treatment and will be randomly assigned to either esketmaine or placebo treatment. Esketamine/placebo will be administered by intranasal route (delivery of medications through the nasal mucosa) two times per week for 4 weeks. Efficacy of the participants will be primarily evaluated through MADRS. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnostic criteria for major depressive disorder
* Participants must have current suicidal ideation with intent
* In the Investigator's opinion, participant must be in need of acute psychiatric hospitalization due to imminent risk of suicide
* Participant has a Montgomery Asberg Depression Rating Scale (MADRS) total score of greater than or equal to (>=) 22 predose on Day 1
* As part of standard of care treatment, participant agrees to be hospitalized voluntarily for a recommended period of 5 days after randomization (that is, through Day 5), and take prescribed non-investigational antidepressant therapy(ies) for at least the duration of the double-blind treatment phase (Day 25)

Exclusion Criteria:

* Participant has a current clinical diagnosis of bipolar or related disorders, intellectual disability, or cluster b personality disorder (example, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, and narcissistic personality disorder)
* Participant meets DSM-IV criteria for borderline personality disorder, based on clinical interview
* Participant has a current or prior diagnosis of a psychotic disorder, major depressive disorder (MDD) with psychosis, or obsessive compulsive disorder
* Participant with a history or current signs and symptoms of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbances
* Participant has uncontrolled hypertension (systolic blood pressure greater than [>] 160 millimeter of mercury [mmHg] or diastolic blood pressure > 90 mmHg) despite diet, exercise or a stable dose of an allowed anti-hypertensive treatment at Screening; or any past history of hypertensive crisis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- United States (14):
  - Birmingham, Alabama
  - San Diego, California
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Towson, Maryland
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208
- [Derived] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- See also: A Double-blind Study to Assess the Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Participants Who are Assessed to be at Imminent Risk for Suicide — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR103162&attachmentIdentifier=197ac6b4-787c-46b2-93a3-5bbc385b3a47&fileName=ESKETINSUI2001_(CR103162)_Additional_Results_Data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received intranasal placebo (1 spray in each nostril at 0, 5 and 10 minutes using 3 devices on a single day) administered twice weekly for 4 weeks on days 1, 4, 8, 11, 15, 18, 22, and 25 along with standard of care antidepressant treatment (determined by the treating physician based on clinical judgment) on Day 1 and continued for the duration of the double-blind treatment phase.
- Esketamine 84 mg: Participants self-administered 1 spray into each nostril (1 spray in each nostril at 0, 5 and 10 minutes using 3 devices on a single day) of Esketamine 84 milligram (mg) twice Weekly for 4 Weeks on Days 1, 4, 8, 11, 15, 18, 22, and Day 25 along with standard of care antidepressant treatment (determined by the treating physician based on clinical judgment) on Day 1 and continued for the duration of the double-blind treatment phase. After Day 1, a single dose reduction from esketamine 84 mg to esketamine 56 mg was permitted if a participant was unable to tolerate the intranasal esketamine 84 mg. Participants continued to receive the reduced dose for the duration of the double-blind treatment phase.
Period: Double Blind (Day 1-25)
Arm/Group | Placebo | Esketamine 84 mg
Started | 32 | 36
Safety | 31 | 35
Completed | 22 (Participants who completed continued to follow-up phase.) | 27 (Participants who completed continued to follow-up phase.)
Not Completed | 10 | 9
Not completed — Adverse Event | 1 | 5
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Period: Follow-Up Phase (Day 26-81)
Arm/Group | Placebo | Esketamine 84 mg
Started | 22 | 27
Completed | 20 | 24
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat Analysis (ITT) analysis set defined as all randomized participants who received at least 1 dose of study medication during the double-blind phase and had both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Esketamine 84 mg | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12.82) | 35.7 (13.4) | 35.8 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 10 | 13 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 1: 4-Hour Post-dose in Montgomery Asberg Depression Rating Scale (MADRS) Total Score (Double-blind Phase)
Description: The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition. The last observation carried forward (LOCF) approach was used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-Predose) to Day 1: 4-hours post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | -9.1 (8.38) | -13.4 (9.03)

2. Secondary Outcome: Percentage of Participants With Sustained Response Based on MADRS Total Score (Double-blind Phase)
Description: Sustained response is defined as a reduction from baseline in MADRS total score of greater than or equal to 50 percent, with onset on Day 1 that is maintained through the end of the double-blind phase (Day 25). The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition. The LOCF approach was used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Day 1 to Day 25
Population: ITT analysis set defined as all randomized participants who received at least 1 dose of study medication during the double-blind phase and had both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Percentage of participants | 6.7 | 11.8

3. Secondary Outcome: Change From Baseline to Day 2 in MADRS Total Score (Double-blind Phase)
Description: The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition. The LOCF approach was used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | -12.8 (9.77) | -19.3 (12.02)

4. Secondary Outcome: Change From Baseline to Double-blind Phase-End Point (Day 25) in MADRS Total Score (Double-blind Phase)
Description: The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition. The LOCF approach was used for missing visit data in the ITT LOCF efficacy analyses. The last post baseline observation was carried forward as the "End Point" for the double-blind phase.
Time Frame: Baseline (Day 1-predose) to Double-blind Phase-End Point (Day 25)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
units on a scale | -23.0 (10.83) | -26.4 (14.52)

5. Secondary Outcome: Percentage of Participants With Response Based on MADRS Total Score During the Double-Blind Phase
Description: Percentage of participants with response (greater than or equal to (>=) 50% improvement from baseline in MADRS total score) during the double- blind phase was assessed. The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition.
Time Frame: Day 1 (4 hours postdose), Day 2 (double blind phase), Double blind phase -Endpoint (Day 25)
Population: ITT analysis set defined as all randomized participants who received at least 1 dose of study medication during the double-blind phase and had both the baseline and the Day 1-4-hour post dose evaluation for the MADRS total score.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Percentage of participants
  Day 1 (4 hours postdose) | 12.9 | 25.7
  Day 2 (double blind phase) | 29.0 | 54.3
  Double blind phase -Endpoint (Day 25) | 54.8 | 74.3

6. Secondary Outcome: Percentage of Participants With Response Based on MADRS Total Score at Follow up Phase Endpoint
Description: Percentage of participants with response (greater than or equal to (>=) 50% improvement from baseline in MADRS total score) during the follow up was assessed. The MADRS consists of 10 items that cover all of the core depressive symptoms (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts). Each item is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptom). A total score (0 to 60) is calculated by adding the scores of all 10 items. For each item as well as the total score, a higher score represents a more severe condition.
Time Frame: Follow up phase-endpoint (Day 81)
Population: The ITT (Follow Up phase) analysis set was defined as all participants who had at least one measurement of MADRS total score during the follow up phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 22 | 27
Percentage of participants | 63.6 | 66.7

7. Secondary Outcome: Change From Baseline to Day 1: 4-hours Post-dose in Suicide Ideation and Behavior Assessment Tool (SIBAT)-Clinical Global Judgment of Suicide Risk (CGJ-SR) Module 8 Score (Double-blind Phase)
Description: SIBAT CGJ-SR: Module 8 operates numerous clinical global impression (CGI) severity scales used in other psychiatric studies. Changes in CGJ-SR designed to categorize clinically meaningful changes in clinician rated suicide risk from 'not at all suicidal' to 'participant is at imminent risk of suicide and immediate need for strong intervention (hospitalization with 24 hour 1:1 observation).' Patient scores for clinician-rated suicide risk: 0 (not suicidal); 1(occasional suicidal ideas, no intervention required);2(some clear suicidal ideas present),3(suicidal risk requires scheduled outpatient follow-up,no immediate intervention),4(suicidal risk requires immediate intervention, no hospitalization). 5( suicidal risk requires immediate hospitalization, no suicide precautions),6 (suicide risk requires hospitalization with suicide precautions). LOCF approach used for missing visit data in ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 1: 4-hours Postdose
Population: ITT analysis set: all randomized participants who received at least 1 dose of study medication during the double-blind phase and had both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score. Here N (overall number of participants analyzed)signifies number of participants who were evaluable for this endpoint.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 33
Units on a scale | 0 [-5 to 1] | 0 [-6 to 1]

8. Secondary Outcome: Change From Baseline to Day 2 in Suicide Ideation and Behavior Assessment Tool (SIBAT)-Clinical Global Judgment of Suicide Risk (SIBAT CGJ-SR) Module 8 Score (Double-blind Phase)
Description: SIBAT CGJ-SR: Module 8 operates like numerous other CGI severity scales used in other psychiatric studies. Changes in CGJ-SR designed to categorize clinically meaningful changes in clinician rated suicide risk from 'not at all suicidal' to 'participant is at imminent risk of suicide and immediate need for strong intervention (hospitalization with 24 hour 1:1 observation).' Patient scores for clinician-rated suicide risk: 0 (not suicidal); 1(occasional suicidal ideas, no intervention required);2(some clear suicidal ideas present),3(suicidal risk requires scheduled outpatient follow-up,no immediate intervention),4(suicidal risk requires immediate intervention, no hospitalization). 5( suicidal risk requires immediate hospitalization, no suicide precautions),6 (suicide risk requires hospitalization with suicide precautions). LOCF approach used for missing visit data in ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 2
Population: ITT analysis set: all randomized participants who received at least 1 dose of study medication during the double-blind phase and had both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | 0 [-6 to 0] | -1.0 [-6 to 1]

9. Secondary Outcome: Change From Baseline to Double-blind Phase-Endpoint (Day 25) Suicide Ideation and Behavior Assessment Tool (SIBAT)-Clinical Global Judgment of Suicide Risk (SIBAT CGJ-SR) Module 8 (Double-blind Phase)
Description: SIBAT CGJ-SR: Module 8 operates like numerous other CGI severity scales used in other psychiatric studies. Changes in CGJ-SR designed to categorize clinically meaningful changes in clinician rated suicide risk from 'not at all suicidal' to 'participant is at imminent risk of suicide and immediate need for strong intervention (hospitalization with 24 hour 1:1 observation).' Patient scores for clinician-rated suicide risk: 0 (not suicidal); 1(occasional suicidal ideas, no intervention required);2(some clear suicidal ideas present),3(suicidal risk requires scheduled outpatient follow-up,no immediate intervention),4(suicidal risk requires immediate intervention, no hospitalization). 5( suicidal risk requires immediate hospitalization, no suicide precautions),6 (suicide risk requires hospitalization with suicide precautions). LOCF approach used for missing visit data in ITT LOCF efficacy analyses. Last post baseline observation was carried forward as "End Point" for the double-blind phase.
Time Frame: Baseline (Day 1-predose) to Double-blind Phase-Endpoint (Day 25)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | -5.0 [-6 to 0] | -5.0 [-6 to 0]

10. Secondary Outcome: Change From Baseline to Follow-up Phase-Endpoint (Day 81) in Suicide Ideation and Behavior Assessment Tool (SIBAT)-Clinical Global Judgment of Suicide Risk Score (Follow-up Phase)
Description: SIBAT CGJ-SR: Module 8 operates like numerous other CGI severity scales used in other psychiatric studies. Changes in CGJ-SR designed to categorize clinically meaningful changes in clinician rated suicide risk from 'not at all suicidal' to 'participant is at imminent risk of suicide and immediate need for strong intervention (hospitalization with 24 hour 1:1 observation).' Patient scores for clinician-rated suicide risk: 0 (not suicidal); 1(occasional suicidal ideas, no intervention required);2(some clear suicidal ideas present),3(suicidal risk requires scheduled outpatient follow-up,no immediate intervention),4(suicidal risk requires immediate intervention, no hospitalization). 5( suicidal risk requires immediate hospitalization, no suicide precautions),6 (suicide risk requires hospitalization with suicide precautions). LOCF approach used for missing visit data in ITT LOCF efficacy analyses. Last post baseline observation was carried forward as "End Point" for follow up phase.
Time Frame: Baseline (Day 1-predose) to Follow-up Phase-Endpoint (Day 81)
Population: as for outcome 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 22 | 27
Units on a scale | -5.0 [-6 to -3] | -5.0 [-6 to -2]

11. Secondary Outcome: Change From Baseline to Day 1: 4- Hours Postdose in SIBAT-Patient-Reported Global Assessment of Suicide Risk (Module 6) Score (Double-blind Phase)
Description: SIBAT was specifically developed to measure rapid change in suicidality, based on concerns that existing scales such as Beck Scale for Suicidal Ideation (BSS) are not designed to discriminate differences associated with rapid change. Patient-rated section includes following modules: Module 1 (M-1)(demographic information,suicide history), M-2(current suicidal thinking),M-3 (protective factors), M-4 (suicide behavior),M-5(suicide risk),M-6(suicide-implicit association test).Patient-reported global assessment of suicide risk summarizes patient's judgment of suicide risk (Module 6). Scores: 0(None), 1(Very weak), 2(Weak), 3(Moderately weak), 4(Mild), 5(Moderate), 6 (Moderately strong), 7(Strong), 8(Extremely strong), 9(Extremely strong,constant). Negative change in score indicates improvement. LOCF approach used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 1: 4-hours postdose
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on scale | -1.0 [-6 to 3] | -1.0 [-7 to 2]

12. Secondary Outcome: Change From Baseline to Day 2 in Suicide Ideation and Behavior Assessment Tool Patient-Reported Global Assessment of Suicide Risk (Module 6) Score (Double-blind Phase)
Description: SIBAT was specifically developed to measure rapid change in suicidality, based on concerns that existing scales such as BSS are not designed to discriminate differences associated with rapid change. Patient-rated section includes following modules: Module 1 (M-1)(demographic information,suicide history), M-2(current suicidal thinking),M-3 (protective factors), M-4 (suicide behavior),M-5(suicide risk),M-6(suicide-implicit association test).Patient-reported global assessment of suicide risk summarizes patient's judgment of suicide risk (Module 6). Scores: 0(None), 1(Very weak), 2(Weak), 3(Moderately weak), 4(Mild), 5(Moderate), 6 (Moderately strong), 7(Strong), 8(Extremely strong), 9(Extremely strong,constant). Negative change in score indicates improvement. LOCF approach used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 2
Population: Intent-To-Treat Analysis (ITT) analysis set defined as all randomized participants who received at least 1 dose of study medication during the double-blind phase and have both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | -1.5 [-7 to 1] | -2 [-8 to 0]

13. Secondary Outcome: Change From Baseline to Double Blind Phase-Endpoint (Day 25) in Suicide Ideation and Behavior Assessment Tool Patient-Reported Global Assessment of Suicide Risk (Module 6) Score (Double-blind Phase)
Description: SIBAT was specifically developed to measure rapid change in suicidality, based on concerns that existing scales such as BSS are not designed to discriminate differences associated with rapid change. Patient-rated section includes following modules: Module 1 (M-1)(demographic information,suicide history), M-2(current suicidal thinking),M-3 (protective factors), M-4 (suicide behavior),M-5(suicide risk),M-6(suicide-implicit association test).Patient-reported global assessment of suicide risk summarizes patient's judgment of suicide risk (Module 6). Scores: 0(None), 1(Very weak), 2(Weak), 3(Moderately weak), 4(Mild), 5(Moderate), 6 (Moderately strong), 7(Strong), 8(Extremely strong), 9(Extremely strong,constant). Negative change in score indicates improvement. LOCF approach used for missing visit data in the ITT LOCF efficacy analyses. Last post baseline observation was carried forward as "End Point" for double-blind phase.
Time Frame: Baseline (Day 1-predose) to Double-blind Phase-Endpoint (Day 25)
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 35
Units on a scale | -3.0 [-9 to 1] | -4.0 [-8 to 0]

14. Secondary Outcome: Change From Baseline to Follow-up Phase-Endpoint (Day 81) in Suicide Ideation and Behavior Assessment Tool Patient-Reported Global Assessment of Suicide Risk (Module 6) Score (Follow-up Phase)
Description: SIBAT was specifically developed to measure rapid change in suicidality, based on concerns that existing scales such as BSS are not designed to discriminate differences associated with rapid change. Patient-rated section includes following modules: Module 1 (M-1)(demographic information,suicide history), M-2(current suicidal thinking),M-3 (protective factors), M-4 (suicide behavior),M-5(suicide risk),M-6(suicide-implicit association test).Patient-reported global assessment of suicide risk summarizes patient's judgment of suicide risk (Module 6). Scores: 0(None), 1(Very weak), 2(Weak), 3(Moderately weak), 4(Mild), 5(Moderate), 6 (Moderately strong), 7(Strong), 8(Extremely strong), 9(Extremely strong,constant). Negative change in score indicates improvement. LOCF approach used for missing visit data in ITT LOCF efficacy analyses, last post baseline observation was carried forward as the "End Point" follow up phase.
Time Frame: Baseline (Day 1-predose) to Follow-up Phase Endpoint (Day 81)
Population: as for outcome 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 22 | 27
Units on a scale | -4.0 [-9 to 0] | -3.0 [-9 to 0]

15. Secondary Outcome: Change From Baseline to Day 1: 4-Hours Postdose in Beck Scale for Suicidal Ideation (BSS) Total Score (Double-blind Phase)
Description: BSS is 21-item self-reported instrument to detect and measure severity of suicidal ideation. BSS measures broad spectrum of attitudes and behaviors associated with risk of suicide. Items in scale assess respondent's suicidal plans, deterrents to suicide, level of openness to revealing suicidal thoughts. First 19 items of scale measure gradations of severity of suicidal wishes,attitude, plans.Statements reflect increasing gradations of this severity,are scored from 0 to 2. Final two items ask about number of suicide attempts, seriousness of intention to die associated with last attempt,they are not used in calculating BSS total score. Total BSS score represents severity of suicide ideation, calculated by summing ratings of first 19 items;total score ranges from 0 to 38, with higher score representing greater suicide ideation. LOCF approach used for missing visit data in ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 1: 4-hours postdose
Population: ITT analysis set: all randomized participants who received at least 1 dose of study medication during the double-blind phase and have both the baseline and the Day 1-4 hour post dose evaluation for the MADRS total score. Here 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 34
Units on a scale | -8.3 (7.12) | -10.2 (9.74)

16. Secondary Outcome: Change From Baseline to Day 2 in Beck Scale for Suicidal Ideation (BSS) Total Score (Double-blind Phase)
Description: BSS is 21-item self-reported instrument to detect and measure severity of suicidal ideation. BSS measures broad spectrum of attitudes and behaviors associated with risk of suicide. Items in scale assess respondent's suicidal plans, deterrents to suicide,level of openness to revealing suicidal thoughts. First 19 items of scale measure gradations of severity of suicidal wishes, attitude, plans.Statements reflect increasing gradations of this severity,are scored from 0 to 2. Final two items ask about number of suicide attempts, seriousness of intention to die associated with last attempt,they are not used in calculating BSS total score. Total BSS score represents severity of suicide ideation, calculated by summing ratings of first 19 items;total score ranges from 0 to 38, with higher score representing greater suicide ideation. LOCF approach used for missing visit data in ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 2
Population: ITT analysis set: all randomized participants who received at least 1 dose of study medication during the double-blind phase and have both the baseline and the Day 1, 4-hour post dose evaluation for the MADRS total score. Here 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 34
Units on a scale | -10.7 (7.73) | -12.9 (9.63)

17. Secondary Outcome: Change From Baseline to Double-blind Phase-Endpoint (Day 25) in Beck Scale for Suicidal Ideation Total Score (Double-blind Phase)
Description: BSS is 21-item self-reported instrument to detect and measure severity of suicidal ideation.BSS measures broad spectrum of attitudes and behaviors associated with risk of suicide. Items in scale assess respondent's suicidal plans, deterrents to suicide, level of openness to revealing suicidal thoughts. First 19 items of scale measure gradations of severity of suicidal wishes, attitude, plans.Statements reflect increasing gradations of this severity,are scored from 0 to 2. Final two items ask about number of suicide attempts, seriousness of intention to die associated with last attempt,they are not used in calculating BSS total score. Total BSS score represents severity of suicide ideation, calculated by summing ratings of first 19 items;total score ranges from 0 to 38, with higher score representing greater suicide ideation. LOCF approach used for missing visit data in ITT LOCF efficacy analyses. Last post baseline observation was carried forward as "End Point" for double-blind phase.
Time Frame: Baseline (Day 1-predose) to Double-blind Phase-endpoint (Day 25)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 31 | 34
Units on a scale | -16.0 (10.54) | -19.3 (9.61)

18. Secondary Outcome: Change From Baseline to Follow-up Phase-Endpoint (Day 81) in Beck Scale for Suicidal Ideation Total Score (Follow-up Phase)
Description: BSS is 21-item self-reported instrument to detect and measure severity of suicidal ideation. BSS measures broad spectrum of attitudes and behaviors associated with risk of suicide. Items in scale assess respondent's suicidal plans, deterrents to suicide, level of openness to revealing suicidal thoughts. First 19 items of scale measure gradations of severity of suicidal wishes, attitude, plans.Statements reflect increasing gradations of this severity,are scored from 0 to 2. Final two items ask about number of suicide attempts, seriousness of intention to die associated with last attempt,they are not used in calculating BSS total score. Total BSS score represents severity of suicide ideation, calculated by summing ratings of first 19 items;total score ranges from 0 to 38, with higher score representing greater suicide ideation. LOCF approach used for missing visit data in ITT LOCF efficacy analyses, last post baseline observation was carried forward as the "End Point" follow up phase.
Time Frame: Baseline (Day 1-predose) to Follow-up Phase-Endpoint (Day 81)
Population: The ITT (Follow Up phase) analysis set was defined as all participants who had at least one measurement of MADRS total score during the follow up phase. Here 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 22 | 26
Units on a scale | -18.0 (9.92) | -20.3 (8.02)

19. Secondary Outcome: Change From Baseline to Day 1: 4-Hours Postdose in Beck Hopelessness Scale (BHS) Total Score (Double-blind Phase)
Description: BHS is paper-based self-reported measure to assess one's level of negative expectations or pessimism regarding future. Consists of 20 true-false items that examine the respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9 are keyed false and 11 are keyed true. Items fall within 3 domains: feelings about future; loss of motivation; future expectations. each response is assigned a score of 0 or 1. Total BHS score is sum of item responses, with range from 0 to 20, with a higher score representing higher level of hopelessness. Total scores that range from 0 to 3 are (normal range), scores 4 to 8 (mild hopelessness, scores 9 to 14 (moderate hopelessness), scores <14 (severe hopelessness). Negative change in score indicates improvement. The LOCF approach was used for missing visit data in the ITT LOCF efficacy analyses.
Time Frame: Baseline (Day 1-predose) to Day 1: 4-hours Postdose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 30 | 35
Units on a scale | -3.1 (5.71) | -4.1 (5.63)

20. Secondary Outcome: Change From Baseline to Double-blind Phase-Endpoint (Day 25) in Beck Hopelessness Scale Total Score (Double-blind Phase)
Description: BHS is paper-based self-reported measure to assess one's level of negative expectations or pessimism regarding future. Consists of 20 true-false items that examine the respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9 are keyed false and 11 are keyed true. Items fall within 3 domains: feelings about future; loss of motivation; future expectations. each response is assigned a score of 0 or 1. Total BHS score is sum of item responses, with range from 0 to 20, with a higher score representing higher level of hopelessness. Total scores that range from 0 to 3 are (normal range), scores 4 to 8 (mild hopelessness, scores 9 to 14 (moderate hopelessness), scores <14 (severe hopelessness). Negative change in score indicates improvement. The LOCF approach was used for missing visit data in the ITT LOCF efficacy analyses. The last post baseline observation was carried forward as the "End Point" for the double-blind phase.
Time Frame: Baseline (Day 1-predose) to Double-blind Phase-Endpoint (Day 25)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Esketamine 84 mg
Number analyzed (Participants) | 30 | 35
Units on a scale | -7.7 (7.81) | -10.3 (5.51)

ADVERSE EVENTS:
Time Frame: Up to Day 81
Description: Safety analysis set included all randomized participants who receive at least 1 dose of study drug in the double-blind phase. Safety (FU) analysis set included all participants who had at least 1 visit during the follow-up phase.
Groups:
- Double Blind (Day 1-25): Placebo: Participants received intranasal placebo (1 spray in each nostril at 0, 5 and 10 minutes using 3 devices on a single day) administered twice weekly for 4 Weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25 along with standard of care antidepressant treatment determined by the treating physician based on clinical judgment on Day 1 and continued for the duration of the double-blind treatment phase.
- Double Blind (Day 1-25): Esketamine 84 mg: Participants self-administered 1 spray into each nostril (1 spray in each nostril at 0, 5 and 10 minutes using 3 devices on a single day) of Esketamine 84 milligram (mg) twice Weekly for 4 Weeks on Days 1, 4, 8, 11, 15, 18, 22, and Day 25 along with standard of care antidepressant treatment determined by the treating physician based on clinical judgment on Day 1 and continued for the duration of the double-blind treatment phase. After Day 1, a single dose reduction from esketamine 84 mg to esketamine 56 mg was permitted if a participant was unable to tolerate the intranasal esketamine 84 mg. Participants continued to receive the reduced dose for the duration of the double-blind treatment phase.
- Follow Up Phase (Day 26-81): Placebo; Follow Up Phase (Day 26-81): Esketamine 84 mg: Participants who completed the double blind treatment phase were continued to follow-up phase for 81 days.
Arm/Group | Double Blind (Day 1-25): Placebo | Double Blind (Day 1-25): Esketamine 84 mg | Follow Up Phase (Day 26-81): Placebo | Follow Up Phase (Day 26-81): Esketamine 84 mg
Serious Adverse Events (participants affected / at risk) | 0/31 | 4/35 | 5/22 | 1/27
Other Adverse Events (participants affected / at risk) | 25/31 | 30/35 | 6/22 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (Day 1-25): Placebo (N=31) | Double Blind (Day 1-25): Esketamine 84 mg (N=35) | Follow Up Phase (Day 26-81): Placebo (N=22) | Follow Up Phase (Day 26-81): Esketamine 84 mg (N=27)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressive Symptom (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 2 | 1 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (Day 1-25): Placebo (N=31) | Double Blind (Day 1-25): Esketamine 84 mg (N=35) | Follow Up Phase (Day 26-81): Placebo (N=22) | Follow Up Phase (Day 26-81): Esketamine 84 mg (N=27)
Hyperacusis (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 4 | 0 | 0
Blepharospasm (Eye disorders) | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 3 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 13 | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 7 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 0 | 0
Feeling Abnormal (General disorders) | 0 | 3 | 0 | 0
Feeling Cold (General disorders) | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1 | 1
Blood Pressure Increased (Investigations) | 0 | 2 | 0 | 0
Weight Increased (Investigations) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 12 | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 5 | 11 | 0 | 1
Headache (Nervous system disorders) | 8 | 11 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 6 | 0 | 0
Sedation (Nervous system disorders) | 2 | 6 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 4 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 6 | 0 | 0
Dissociation (Psychiatric disorders) | 4 | 11 | 0 | 0
Euphoric Mood (Psychiatric disorders) | 2 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 3
Panic Attack (Psychiatric disorders) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Intranasal Paraesthesia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.